CLINICAL TRIAL: NCT00497367
Title: A Prospective, Single-arm, Multicenter 2-phase Feasibility Study to Assess the TAXUS Petal Paclitaxel-Eluting Bifurcation Coronary Stent System (TAXUS Petal)for the Treatment of de Novo Atherosclerotic Bifurcation Lesions
Brief Title: Safety Study to Assess the Feasibility of Use in Humans of the TAXUS Petal Bifurcation Coronary Stent System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: S2030; S2030-FHU-2007
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Diseases
Keywords: safety; feasibility; bifurcation; lesion; de novo; intervention
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAXUS® Petal™ Paclitaxel-Eluting Coronary Stent (Experimental): This arm received the TAXUS® Petal™ Paclitaxel-Eluting Coronary Stent.
  Interventions: Device: Percutaneous Coronary Intervention (PCI) TAXUS Petal

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (PCI) TAXUS Petal — TAXUS Petal, paclitaxel eluting stent

SUMMARY:
The purpose of this study is to determine the safety and feasibility of use in humans of the TAXUS Petal Paclitaxel-Eluting Bifurcation Coronary Stent System in the treatment of de novo lesions in native coronary arteries involving a major side branch. The TAXUS® Petal™ is an investigational device with an indication of improving coronary artery luminal diameter while maintaining side branch access in subjects with symptomatic ischemic disease due to discrete atherosclerotic bifurcation lesions

DETAILED DESCRIPTION:
To assess the safety and feasibility of use in humans of the TAXUS Petal Paclitaxel-Eluting Bifurcation Coronary Stent System (TAXUS® Petal™) for the treatment of de novo atherosclerotic bifurcation lesions (by visual estimate):

* Phase 1:

  * Main branch: 3.0 to 3.5 mm RVD and lesion length ≤20 mm
  * Side branch: 2.5 to 3.5 mm RVD and lesion length ≤14 mm
* Phase 2:

  * Main branch: 3.0 to 3.5 mm RVD and lesion length ≤28 mm
  * Side branch: 2.25 to 3.5 mm RVD and lesion length ≤14 mm

Bifurcation main branch (MB) lesion length will be measured from the proximal shoulder of the most proximal lesion to the distal shoulder of the most distal lesion. Bifurcation side branch (SB) lesion length will be measured from the proximal shoulder of the side branch (if the ostium is disease-free) or the side branch ostium (if the disease continues into the main branch) to the distal side branch shoulder of the most distal lesion. At follow-up, the entire stented region will be used to determine MLD and %DS.

ELIGIBILITY:
Inclusion Criteria - Phases 1 and 2

* Age is ≥18 years old and ≤80 years old
* Eligible for PCI
* Acceptable candidate for CABG
* Documented stable angina pectoris (CCS Classification 1, 2, 3, or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* LVEF known to be ≥40%
* Clinical angiographic success in non-target lesion (if a non-target lesion is treated)
* Subject (or legal guardian) understands the study requirements and procedures and provides written Informed Consent before any study tests or procedures are performed
* Subject willing to comply with follow-up evaluations

Exclusion Criteria - Phases 1 and 2

* Contraindication to ASA, or to Thienopyridine derivatives (e.g. Clopidogrel, Ticlopidine)
* High risk of bleeding
* Known hypersensitivity to paclitaxel
* Known allergy to stainless steel
* Known allergy to platinum
* Previous treatment of the target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent
* Previous treatment of the target vessel with BMS within 9 months before index procedure
* Previous treatment of any non-target vessel with any anti-restenotic drug-coated or DES within 9 months before index procedure
* Previous treatment with intravascular brachytherapy in the target vessel
* Planned PCI or CABG post-index procedure
* Planned target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter
* Documented MI within 72 hours prior to index procedure
* CK > 2 x ULN + positive CK-MB OR
* CK > 2 x ULN + positive troponin OR
* If no CK-MB or troponin was drawn, patients are excluded with CK > 2xULN
* As per protocol definitions found in Appendix A:
* CVA within the past 6 months
* Cardiogenic shock
* Acute or chronic renal dysfunction
* Prior anaphylactic reaction to contrast agents
* Leukopenia
* Thrombocytopenia
* Thrombocytosis
* Active peptic ulcer or active GI bleeding
* Current treatment, or past-treatment within 12 months of the index procedure, with paclitaxel or other chemotherapeutic agents
* Anticipated treatment with paclitaxel or oral rapamycin within 9 months of index procedure
* Subject's (men and women) known intention to procreate within 9 months of index procedure
* Positive pregnancy test or nursing an infant within 7 days prior to index procedure
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit subject's ability to comply with study follow-up or impact study scientific integrity
* Currently participating in another investigational drug or device clinical study
* Planned surgery at time of enrollment within the next 9 months after index procedure

Angiographic Inclusion Criteria - Phases 1 & 2

* Target Lesion (main and / or side branch):
* located in native coronary artery
* must be de novo
* main branch %DS is ≥50% and <100%
* is a bifurcation lesion with an angle ≥30º and ≤90º
* is enrolled after successful pre-dilatation of the target vessel

Angiographic Inclusion Criteria - Phase 1

* Main branch of target lesion located in parent branch of LAD or LCx or RCA
* Target lesion located in proximal or mid-section of vessel only (crux of RCA [distal RCA] is allowed)
* Main branch RVD ≥3.00 mm to ≤3.5 mm; lesion length ≤20 mm (to be covered by TAXUS® Petal™ stent and maximum of 1 additional TAXUS stent ≤12 mm in length)
* Side branch RVD ≥2.5 mm to ≤3.5 mm; lesion length ≤14 mm to be treated by maximum of 1 TAXUS stent ≤16 mm in length Angiographic Inclusion Criteria - Phase 2
* Main branch of target lesion located in parent branch of LAD or LCx or RCA without restrictions
* Main branch RVD ≥3.00 mm to ≤3.5 mm; lesion length ≤28 mm (to be covered by TAXUS® Petal™ stent and maximum of 1 additional TAXUS stent ≤20 mm in length)
* Side branch RVD ≥2.25 mm to ≤3.5 mm; lesion length ≤14 mm to be treated by maximum of 1 TAXUS stent ≤16 mm in length

Angiographic Exclusion Criteria - Phases 1 & 2

* Target lesion located in left main (protected or unprotected)
* Medina Classification 0.0.1
* Target lesion is restenotic
* Target lesion located in a SVG or mammary artery graft
* Target lesion accessed via SVG or mammary artery graft
* Target lesion is <5 mm from BMS
* Target lesion is <5 mm from second side branch vessel ≥1.5 mm in diameter
* Untreated lesions with ≥50% DS or thought to impair flow remaining in target vessel
* Target lesion and/or vessel proximal to target lesion moderately or severely calcified
* Target lesion and/or target vessel proximal to target lesion severely tortuous
* Main branch target lesion located within or distal to a >60° bend in target vessel
* Target vessel with angiographic presence of probable or definite thrombus
* Unprotected LM disease
* Protected LM disease with target lesion in LAD or LCx (subject may be enrolled if only lesion is target lesion in RCA)

Angiographic Exclusion Criteria

* Phase 1: Target lesion TIMI flow <3
* Phase 2: Target lesion TIMI flow <2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Composite safety endpoint at 30 days post-procedure: • All-cause mortality • Documented myocardial infarction • TVR | 30 days

SECONDARY OUTCOMES:
Device Success Technical Success Clinical Procedural Success Device malfunctions Ease-of-Use parameters Clinical endpoints Main branch and side branch angiographic endpoints Main branch and side branch IVUS endpoints | Index procedure, 30 days, 6 months and 1 - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Ormiston, MD, Principal Investigator — Auckland City Hospital, Grafton, Auckland NZ
Locations (4):
- Institut Hospitalier Jacques Cartier-ICPS, 6, Avenue du Noyer Lambert, Massy, France
- HELIOS Klinikum Siegburg, Ringstrasse 49, Siegburg, Germany
- New Zealand (2):
  - Mercy Angiography Unit, 98 Mountain Road, First Floor, Auckland, Epsom
  - Auckland City Hospital, Cardiac Investigations Unit, Park Road, Auckland, Grafton

REFERENCES:
- [Derived] Ormiston JA, Lefevre T, Grube E, Allocco DJ, Dawkins KD. First human use of the TAXUS Petal paclitaxel-eluting bifurcation stent. EuroIntervention. 2010 May;6(1):46-53. PMID 20542797